CLINICAL TRIAL: NCT00004490
Title: Phase III Randomized Study of Sodium Dichloroacetate in Children With Congenital Lactic Acidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14271; UF-G-FDR001500; UF-G-183-92
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Lactic Acidosis
Keywords: disease-related problem/condition; inborn errors of metabolism; lactic acidosis; quality of life; rare disease
MeSH Terms: conditions — Acidosis, Lactic; Metabolism, Inborn Errors; Rare Diseases | interventions — Dichloroacetic Acid

INTERVENTIONS:
Drug: sodium dichloroacetate

SUMMARY:
OBJECTIVES:

I. Compare the safety of sodium dichloroacetate (DCA) vs placebo in children with congenital lactic acidosis.

II. Determine the quality of life of these patients.

III. Determine the pharmacokinetics and metabolic fate of DCA over the course of drug administration in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, crossover study. Patients are stratified according to age (3 months to 2 years vs over 2 to 18 years).

All patients receive at least 12 months of sodium dichloroacetate (DCA) during a 2 year period of double blind, crossover evaluation of DCA and placebo by mouth.

Quality of life is assessed before treatment and periodically during treatment.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of congenital lactic acidosis (CLA) meeting the following criteria: Three basal venous lactates at least 2.5 mM, arterial lactates at least 2.0 mM, or CSF lactates at least 2.5 mM OR any combination of these, obtained over at least 1 month and within 6 months OR Increase in blood lactate at least 1.0 mM over basal following a carbohydrate meal challenge

AND

Enzymatic or molecular genetic proof of a defect of pyruvate dehydrogenase complex, one or more respiratory chain enzymes, or a Krebs cycle enzyme OR Over production of C14-lactate from C14-glucose by cultured skin fibroblasts

AND

Ability to withstand an 8 hour (if 2 years and under) or 12 hour (if over 2 years) fast without developing hypoglycemia (blood glucose less than 50 mg/dL)

No secondary lactic acidosis due to impaired oxygenation or circulation

No hyperlactatemia associated with proven biotinidase deficiency (biotin responsive CLA) or with enzyme deficiencies of gluconeogenesis

No primary, defined organic acidurias other than lactic acidosis, for which effective therapy is available (e.g., propionic aciduria)

No primary disorders of amino acid metabolism or fatty acid oxidation

No malabsorption syndromes associated with D-lactic acidosis

--Prior/Concurrent Therapy--

No chronic dialysis

--Patient Characteristics--

Hepatic: No primary hepatic disease unrelated to CLA

Renal: Creatinine less than 1.2 mg/dL OR Creatinine clearance at least 60 mL/min

Other: No concurrent infection or fever

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45
Dates: Start 1998-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Stacpoole, Study Chair — University of Florida